CLINICAL TRIAL: NCT02987907
Title: The Impact on Therapeutic Effect and Tolerance of Treatment for Patients With Hepatocellular Carcinoma in Transcatheter Arterial Chemoembolization (TACE) of Dexamethasone Application: A Random, Double-blind, Controlled, Clinical Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Shaohua, Attending Doctor, Department of Hepatobiliary Pancreatic Surgery, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2016-024-01
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment group (Experimental): use dexamethasone 10mg (2ml) I.A. during TACE
  Interventions: Drug: Dexamethasone
- control group (Placebo Comparator): use normal saline 2ml I.A. during TACE
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — use dexamethasone 10mg (2ml) I.A. during TACE
  Arms: treatment group
Drug: Normal Saline — use normal saline 2ml I.A. during TACE
  Arms: control group

SUMMARY:
The current random, double-blind, controlled, clinical trial was designed to evaluate the impact on therapeutic effect and tolerance of treatment for patients with hepatocelluclar carcinoma in transcatheter arterial chemoembolization (TACE) of dexamethasone application.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old;
* ECOG PS<3;
* proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
* meeting at least 1/4: 1) multiple nodules, 2) single tumor but not suitable for resection, 3) vascular invasion exists, 4) distant metastasis excluding CNS and bone
* not previous treated for tumor;
* Child-Pugh A or B;
* at least one measurable lesion according mRECIST;
* cannot afford sorafenib;
* the lab test could meet: neutrophil count≥1.5×109/L; hemoglobin≥80g/L; platelet count≥60×109/L; serum albumin≥28g/L; total bilirubin<3-times upper limit of normal; ALT<5-times upper limit of normal; AST<5-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 6 seconds; INR≤2.3
* sign up consent;
* unrolled by other clinical trials about hepatocellular carcinoma.

Exclusion Criteria:

* cannot tolerate TACE;
* CNS or bone metastasis exits;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrage or cardiac/brain vascular events within 30 days;
* pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
response rate (RR) | 1 month after TACE
proportions of participants with severe adverse events according to CTCAE v4.03 | 1 month after TACE

SECONDARY OUTCOMES:
overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
time to progression (TTP) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided